CLINICAL TRIAL: NCT02796170
Title: Inhibition of Urinary Angiotensinogen and the Reduction of Blood Pressure by SGLT2 Inhibition in Patients With Type 2 Diabetes
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Tulane University School of Medicine (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Organization: Tulane University (Other)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 812701
Record Dates: First submitted 2016-04-26; First posted 2016-06-10 (Estimated); Results first posted 2022-11-01 (Actual); Last update posted 2022-11-01 (Actual); Status verified 2022-10

CONDITIONS: Type 2 Diabetes; Hypertension
Keywords: SGLT-2 inhibitor; urinary angiotensinogen
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Hypertension | interventions — dapagliflozin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dapagliflozin (Active Comparator): Participants underwent 6 weeks of Dapagliflozin or placebo (washout period for 2 weeks) and then crossed over to 6 weeks of placebo or Dapagliflozin.
  Interventions: Drug: Dapagliflozin; Drug: Placebo
- Placebo (Active Comparator): Participants underwent 6 weeks of Dapagliflozin or placebo (washout period for 2 weeks) and then crossed over to 6 weeks of placebo or Dapagliflozin.
  Interventions: Drug: Dapagliflozin; Drug: Placebo

INTERVENTIONS:
Drug: Dapagliflozin — 5mg pill taken once daily
Drug: Placebo — 5mg pill taken once daily- placebo of Dapagliflozin

SUMMARY:
To assess the effect of sodium-glucose cotransporter 2 (SGLT-2) inhibitors on blood pressure and urinary angiotensinogen. This is a cross over study design, where 40 subjects will receive Dapagliflozin for 6 weeks followed by placebo for 6 weeks, or placebo for 6 weeks followed by Dapagliflozin for 6 weeks. In addition there will be an arm of 10 subjects who will receive sulfonylurea in an open label as a comparative to the cross over subjects to assess if the effect of Dapagliflozin may also be in part due to improved glycemic control.

DETAILED DESCRIPTION:
Clinical trials of two SGLT2 inhibitors, canagliflozin and dapagliflozin, have reported drops in systolic blood pressure of ~5 mmHg. Inappropriate activation of intrarenal renin-angiotensin system (RAS) is a major contributor to the increased arterial pressure and tissue injury including diabetic nephropathy. A key factor in the intrarenal RAS activation is stimulation of intrarenal angiotensinogen (AGT) which is the precursor of angiotensin peptides. From previous studies, it has been shown that high blood sugars in patients with type1 and type 2 diabetes mellitus is accompanied by elevated intrarenal AGT and urinary AGT levels. High glucose results in stimulation of AGT production. The high glucose levels augments intrarenal AGT levels in diabetes mellitus leading to the development of high blood pressure and diabetic nephropathy.

The investigators propose to conduct a single-center randomized, double blind, cross over study of the effect of Dapagliflozin over 6 weeks, followed by placebo over 6 weeks on the other treatment allocation (those getting placebo first will cross over to Dapagliflozin and vice versa). Treatment will be stratified according to the underlying presence or absence of hypertension.

1. Type 2 diabetes with hypertension and on renin-angiotensin-aldosterone system (RAAS) blocking drugs with stable blood pressure on therapy; n= 20
2. Type 2 diabetes without hypertension and not on RAAS blocking drugs n=10

If unable to recruit 10 participants without hypertension the investigators will increase the number with hypertension for a total of 30. Stratification by hypertension status will remain and is important in understanding the effect of SGLT2 inhibition in patients not on BP lowering drugs.

In addition a Sulfonylurea (SU) arm will also be included - 10 participants who are on metformin and other background therapy (with the exclusion of SGLT-2 inhibitor and sulfonylurea) will be recruited. This will be an open-labeled arm. Participants will assessed at baseline. Participants will then receive usual care for 6 weeks. At the end of 6 weeks, participants will then undergo another assessment before being provided SU for 6 weeks. At the end of 6 weeks, participants will undergo assessment again. The aim is to determine whether any effects seen with Dapagliflozin are specific to that drug or related simply to improved glycemic control.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes with hypertension and on RAAS blocking drugs OR
* Type 2 diabetes without hypertension and not on RAAS blocking drugs
* Hemoglobin A1c between 7% and 9% (inclusive)
* Estimated glomerular filtration rate (eGFR) ≥60 ml/min
* Capacity to understand and sign informed consent

Exclusion Criteria:

* Severe hepatic insufficiency and/or significant abnormal liver function defined as aspartate aminotransferase (AST) and/or alanine aminotransferase (ALT) >3x upper limit of normal (ULN)
* Total bilirubin >2.0 mg/dL
* Positive serologic evidence of current infectious liver disease, including Hepatitis B viral antibody immunoglobulin M (IGM), Hepatitis B surface antigen, and Hepatitis C virus antibody
* Estimated glomerular filtration rate (eGFR) <60 ml/min
* Recent cardiovascular events with the last 2 months: acute coronary syndrome (ACS), hospitalization for unstable angina or acute myocardial infarction, acute stroke or transient ischemic attack (TIA), or post coronary artery revascularization
* Congestive Heart Failure defined as New York Heart Association (NYHA) class IV, unstable or acute congestive heart failure
* Pregnant or breastfeeding patients
* Patients who, in the judgement of the investigator, may be at risk for dehydration
* Blood pressure at enrollment: Systolic ≥165 mmHg and/or Diastolic ≥110 mmHg; At randomization: Systolic ≥160 mmHg and/or Diastolic ≥100 mmHg
* Use of SGLT-2 inhibitor class drugs is an exclusion for all patients. For patients in the sulfonylurea arm, use of sulfonylurea class drugs is an exclusion.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2019-08 (Actual); Study Completion 2020-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dragana Lovre, MD, Principal Investigator — Tulane University School of Medicine; Tina Thethi, MD, Principal Investigator — AdventHealth
Locations (1):
- Tulane University, New Orleans, Louisiana, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Dapagliflozin First Then Placebo: Participants underwent 6 weeks of Dapagliflozin (washout period for 2 weeks) and then crossed over to 6 weeks of placebo.
  Dapagliflozin: 5mg pill taken once daily
  Placebo: 5mg pill taken once daily.
- Placebo First Then Dapagliflozin: Participants underwent 6 weeks of placebo (washout period for 2 weeks) and then crossed over to 6 weeks of Dapagliflozin.
  Placebo: 5mg pill taken once daily Dapagliflozin: 5mg pill taken once daily
Period: Overall Study
Arm/Group | Dapagliflozin First Then Placebo | Placebo First Then Dapagliflozin
Started | 8 | 3
Completed | 5 | 3
Not Completed | 3 | 0
Not completed — Lost to Follow-up | 3 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dapagliflozin First Then Placebo | Placebo First Then Dapagliflozin | Total
Number analyzed (Participants) | 8 | 3 | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 7 | 3 | 10
  >=65 years | 1 | 0 | 1
Age, Continuous [Mean (Standard Deviation); unit: Years] | 56.5 (7.8) | 52.7 (6.7) | 55.5 (7.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 1 | 8
  Male | 1 | 2 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 2 | 6
  White | 3 | 0 | 3
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 8 | 3 | 11
Weight [Mean (Standard Deviation); unit: Kg] | 89.3 (17.6) | 114.5 (14.9) | 96.2 (20.0)
BMI [Mean (Standard Deviation); unit: Kg/m^2] | 32.6 (7.4) | 38.2 (8.4) | 34.1 (7.7)
HbA1c [Mean (Standard Deviation); unit: HbA1c %] | 8.0 (1.3) | 7.9 (0.8) | 8.0 (1.1)
Average Systolic Blood pressure [Mean (Standard Deviation); unit: mmHg] | 119.0 (8.5) | 121.3 (19.1) | 119.6 (11.2)
Average Diastolic blood pressure [Mean (Standard Deviation); unit: mmHg] | 74.0 (4.1) | 79.3 (7.1) | 75.4 (5.3)
Average Heart Rate [Mean (Standard Deviation); unit: bpm] | 83.1 (10.9) | 76.5 (13.3) | 81.3 (11.3)
Total Cholesterol [Mean (Standard Deviation); unit: mg/dL] | 175.4 (43.8) | 141.3 (11.4) | 166.1 (40.3)
HDL Cholesterol [Mean (Standard Deviation); unit: mg/dL] | 55.3 (17.6) | 43.3 (4.0) | 52.0 (15.8)
Triglycerides [Mean (Standard Deviation); unit: mg/dL] | 192.8 (184.5) | 111.0 (57.4) | 170.5 (161.1)
LDL Cholesterol [Mean (Standard Deviation); unit: mg/dL] | 80.6 (15.5) | 78.3 (8.4) | 79.9 (13.3)
Estimated glomerular filtration rate (eGFR) [Mean (Standard Deviation); unit: mL/min/1.73m2] | 93.0 (15.4) | 89.0 (5.6) | 91.9 (13.3)
B-blockers [Count of Participants; unit: Participants] | 2 | 1 | 3
Calcium antagonists [Count of Participants; unit: Participants] | 2 | 1 | 3
angiotensin converting enzyme (ACE)-I/ angiotensin receptor blocker (ARB) [Count of Participants; unit: Participants] | 6 | 3 | 9
Statins [Count of Participants; unit: Participants] | 7 | 3 | 10
Diuretics [Count of Participants; unit: Participants] | 3 | 2 | 5
Metformin [Count of Participants; unit: Participants] | 8 | 3 | 11
Sulfonylurea [Count of Participants; unit: Participants] | 2 | 1 | 3
Glucagon-like peptide-1 (GLP-1)/Dipeptidyl Peptidase-4 (DPP-4) [Count of Participants; unit: Participants] | 2 | 1 | 3
Insulin [Count of Participants; unit: Participants] | 3 | 0 | 3

OUTCOME MEASURES:

1. Primary Outcome: Change in Blood Pressure From Baseline to 6 Weeks Measured by ABPM
Description: Blood pressure was measured at baseline with a 24 hour ambulatory blood pressure machine (ABPM), and again after 6 weeks of treatment.
Time Frame: Baseline to 6 weeks
Population: Out of the 8 participants who completed the study, 5 Participants had full data analyzed for this outcome measure, where three participants had the ABPM missing, so they were excluded from the final data analysis.
Measure: Mean (Standard Deviation); unit: mmHg
Groups:
- Placebo: Placebo: 5mg pill taken once daily
Arm/Group | Dapagliflozin | Placebo
Number analyzed (Participants) | 5 | 5
mmHg
  Systolic Blood pressure | -10.72 (6.17) | 1.94 (17.01)
  Diastolic blood pressure | -3.34 (4.2) | 1.56 (15.05)

2. Secondary Outcome: Change in Urinary AGT Levels From Baseline to 6 Weeks
Description: Urinary Angiotensinogen (AGT) was measured through the collection of 24 hour urine at baseline and again after 6 weeks of treatment. Angiotensinogen was normalized to creatinine.
Time Frame: Baseline to 6 weeks
Population: Out of the 8 participants who completed the study, 5 Participants had full data analyzed for this outcome measure, where three participants had the AGT data missing, so they were excluded from the final data analysis.
Measure: Mean (Standard Deviation); unit: ng/mg
Arm/Group | Dapagliflozin | Placebo
Number analyzed (Participants) | 5 | 5
ng/mg | 53.85 (98.79) | 39.69 (58.37)

ADVERSE EVENTS:
Time Frame: Each participant was assessed for adverse events in the duration of 16 weeks
Arm/Group | Dapagliflozin | Placebo
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/3
Other Adverse Events (participants affected / at risk) | 0/8 | 0/3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-06-20): https://cdn.clinicaltrials.gov/large-docs/70/NCT02796170/Prot_SAP_000.pdf